CLINICAL TRIAL: NCT03686215
Title: Pivotal Study of the LUM Imaging System for Assisting Intraoperative Detection of Residual Cancer in the Tumor Bed of Female Patients With Breast Cancer
Brief Title: Investigation of Novel Surgical Imaging for Tumor Excision
Acronym: INSITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lumicell, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL0007; 5R44CA211013-02 (NIH)
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: breast cancer surgery; lumpectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive the device intervention. All subjects will receive the study drug.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking will only be applied until the standard of care surgery is complete. At time of randomization, the study arm will be revealed to the study team. The pathologist will be masked to the type of tissue obtained from the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device Intervention: LUM Imaging System used during surgery (Experimental): The LUM Imaging Device will be used to look inside the lumpectomy cavity to see if the dye indicates any areas that may contain residual tumor. If the imaging identifies that there may be cancer cells remaining in the lumpectomy cavity, the surgeon will remove an additional piece of tissue. This process will be continued until a negative reading from the device is obtained or a maximum of 2 shaves of additional tissue has been removed. Patients in this arm will receive the study drug, LUM015.
  Interventions: Combination Product: Study Device Arm
- Standard of Care Arm (No Intervention): The LUM Imaging Device will not be used to guide additional tissue removal. Patients in this arm will receive the study drug, LUM015.

INTERVENTIONS:
Combination Product: Study Device Arm — LUM015 will be administered 2 to 6 hours prior to surgery. The LUM Imaging device will be used to assist in the removal of additional tumor tissue.
  Other Names: LUM Imaging System
  Arms: Device Intervention: LUM Imaging System used during surgery

SUMMARY:
This is a multi-center, two-arm randomized, blinded pivotal study to demonstrate the safety and efficacy of the LUM Imaging System (LUM015 imaging agent in conjunction with the LUM Imaging Device and decision software), in identifying residual cancer in the lumpectomy bed of female breast cancer patients undergoing breast surgery in order to assist surgeons in reducing the rates of positive margins.

All enrolled subjects will be injected with LUM015 prior to surgery. Surgeons are blinded to whether a participant will be randomized into the device arm until after the standard of care lumpectomy is complete. Participants will then be randomized to receiving the device. Therapeutic (LUM guided) shaves will be removed based on the guidance of the LUM Imaging System. Patients will be followed until their first standard of care post-operative follow-up visit.

DETAILED DESCRIPTION:
All subjects will be injected with LUM015. The injection of the study drug will occur 2-6 hours prior to surgery at a dose of 1.0 mg/kg. Surgeons will complete the standard of care lumpectomy. Prior to removing any shaves as part of the standard of care, the surgeon will use the LUM Imaging System to scan and image the cavity where shaves will be obtained. The system will not provide guidance. The intent of the standard of care lumpectomy procedure is to achieve negative margins.

Randomization of whether the patient will receive the device will be revealed after the completion of the standard of care lumpectomy. If the patient is randomized to the non-device arm, then the surgeon will complete the surgery per their standard practice. If the patient is randomized to the device arm, the surgeon will use the LUM Imaging Device to scan inside the lumpectomy cavity to indicate areas that may contain residual tumor. If the imaging system identifies that there may be cancer cells remaining in the lumpectomy cavity, the surgeon will remove an additional piece of tissue. This process will be continued until a negative reading from the device is obtained or a maximum of 2 shaves of additional tissue has been removed in each orientation.

Study treatment ends when the surgery is completed. All patients will continue their enrollment in the study until their first follow-up visit and they will continue to be followed until the medical team determines no further surgical intervention is required. Patients who have consented to completing Quality of Life Questionnaires will be in the study until the schedule of questionnaires is complete. Patients with adverse events that are determined to be possibly related to the LUM Imaging System will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed primary invasive breast cancer, ductal carcinoma in situ (DCIS) or primary invasive breast cancer with a DCIS component.
* Female, age of 18 years or older.
* Subjects must be scheduled for a lumpectomy for a breast malignancy.
* Subjects must be able and willing to follow study procedures and instructions.
* Subjects must have received and signed an informed consent form.
* Subjects must have no uncontrolled serious medical problems except for the diagnosis of breast cancer, as per the exclusion criteria listed below.
* Subjects must have organ and marrow function within limits as defined below:

  * Leukocytes > 3,000/microlitre (mcL).
  * Platelets > 75,000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST (SGOT))/alanine transaminase (ALT (SGPT)) < 2.5 X institutional upper limit of normal
  * Creatinine ≤ 1.5 mg/dL or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Subjects who have been diagnosed with bilateral breast cancer and are undergoing bilateral resection procedure
* Subjects who are pregnant. Breastfeeding should be discontinued if the mothers is treated with Pegulicianine (LUM015)
* Subjects who are sexually active and not willing/able to use 2 medically acceptable forms of contraception (hormonal or barrier method of birth control, abstinence) upon entering the study and for 60 days after injection of LUM015.
* Subjects who have taken an investigational drug within 30 days of enrollment.
* Subjects who will have administration of methylene blue or any dye for sentinel lymph node mapping on the day of the surgery prior to imaging the lumpectomy cavity with the LUM Imaging Device.
* Subjects who have not recovered from adverse events due to other pharmaceutical or diagnostic agents.
* Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 110 mm Hg; those subjects with known hypertension (HTN) should be stable with controlled HTN while under pharmaceutical therapy.
* History of allergic reaction to polyethylene glycol (PEG).
* History of allergic reaction to any oral or intravenous contrast agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, chronic obstructive pulmonary disease (COPD) or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive individuals on combination antiretroviral therapy are ineligible.
* Any subject for whom the investigator feels participation is not in the best interest of the subject.
* Subjects undergoing a second lumpectomy procedure because of positive margins in a previous surgery prior to entering this study
* Subjects with post-biopsy hematomas greater or equal to 2 cm that are visible on physical exam or detected during pre-operative observations.
* Subjects with prior ipsilateral breast cancer surgeries, mastectomies, breast reconstructions or implants.s with prior ipsilateral breast cancer surgeries, mastectomies, breast reconstructions or implants
* Subjects with prior ipsilateral reduction mammoplasties (breast reductions) performed less than 2 years prior to enrollment to this study.
* Subjects previously treated with systemic therapies to treat the cancer to be removed during this clinical investigation, such as neo-adjuvant chemotherapy or hormonal therapy.
* Subjects undergoing breast conserving surgery whose resected specimen (main lump, shaves, or any other resected tissue) will be evaluated with frozen section after the LUM-guided removal of shaves.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Smith, MD, PhD, Principal Investigator — Massachusetts General Hospital; Jorge Ferrer, PhD, Study Director — Lumicell, Inc.
Locations (14):
- United States (14):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Stanford Hospital and Clinics, Palo Alto, California
  - Morton Plant Mease Health Care Oncology Research, Clearwater, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Comprehensive Breast Care Center/Beaumont Health, Royal Oak, Michigan
  - Duke Cancer Center, Durham, North Carolina
  - Novant Health Salem Surgical Associates, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - CHI Franciscan Research Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith BL, Hunt KK, Carr D, Blumencranz PW, Hwang ES, Gadd MA, Stone K, Dyess DL, Dodge D, Valente S, Dekhne N, Clark P, Lee MC, Samiian L, Lesnikoski BA, Clark L, Smith KP, Chang M, Harris DK, Schlossberg B, Ferrer J, Wapnir IL. Intraoperative Fluorescence Guidance for Breast Cancer Lumpectomy Surgery. NEJM Evid. 2023 Jul;2(7):EVIDoa2200333. doi: 10.1056/EVIDoa2200333. Epub 2023 Apr 27. PMID 38320161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 406 injected with LUM015 (LUMISIGHT), 14 withdrawn before randomization.
Groups:
- Device Intervention: Lum Imaging Device Used During Surgery: The LUM Imaging Device was used to examine inside the lumpectomy cavity to determine if the dye indicated any areas that might contain residual tumor. If the imaging tested positive for the cancer cells remaining in the lumpectomy cavity, the surgeon would remove an additional piece of tissue. This process was continued until a negative reading from the device was obtained or a maximum of 2 shaves of additional tissue had been removed. Patients in this arm received the study drug, LUM015.
  Study Device Arm: LUM015 was administered 2 to 6 hours prior to surgery. The LUM Imaging device was used to assist in the removal of additional tumor tissue.
- Standard of Care Arm: The LUM Imaging Device was not used to guide additional tissue removal. Patients in this arm received the study drug, LUM015.
- Withdrawn Before Randomization: All the patients injected with LUM015 but withdrawn before randomization after standard of care.
Period: Overall Study
Arm/Group | Device Intervention: Lum Imaging Device Used During Surgery | Standard of Care Arm | Withdrawn Before Randomization
Started | 357 | 35 | 14
Completed | 356 | 35 | 0
Not Completed | 1 | 0 | 14
Not completed — Adverse Event | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 4
Not completed — Device issue | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Device Intervention: LUM Imaging System Used During Surgery: The LUM Imaging Device was used to examine inside the lumpectomy cavity to determine if the dye indicated any areas that might contain residual tumor. If the imaging tested positive for the cancer cells remaining in the lumpectomy cavity, the surgeon would remove an additional piece of tissue. This process was continued until a negative reading from the device was obtained or a maximum of 2 shaves of additional tissue had been removed. Patients in this arm received the study drug, LUM015.
  Study Device Arm: LUM015 was administered 2 to 6 hours prior to surgery. The LUM Imaging device was used to assist in the removal of additional tumor tissue.
- Withdrawn Before Randomization: All the patients injected with LUM015 but withdrawn before randomization.
- Total: Total of all reporting groups
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery | Standard of Care Arm | Withdrawn Before Randomization | Total
Number analyzed (Participants) | 357 | 35 | 14 | 406
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 184 | 19 | 8 | 211
  >=65 years | 173 | 16 | 6 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (9.6) | 61.6 (9.9) | 61.6 (11.6) | 62.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357 | 35 | 14 | 406
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 0 | 12
  Not Hispanic or Latino | 336 | 34 | 13 | 383
  Unknown or Not Reported | 10 | 0 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 21 | 1 | 0 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 22 | 4 | 0 | 26
  White | 297 | 27 | 13 | 337
  More than one race | 4 | 0 | 0 | 4
  Unknown or Not Reported | 12 | 2 | 1 | 15
Region of Enrollment [Number; unit: participants]
  United States | 357 | 35 | 14 | 406
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (6.7) | 31.0 (5.9) | 29.8 (6.8) | 29.9 (6.6)
Menopausal Status [Count of Participants; unit: Participants]
  Post | 299 | 28 | 12 | 339
  Pre/Peri | 58 | 7 | 2 | 67
Mammographic breast density [Count of Participants; unit: Participants]
  Almost Entirely Fatty | 5 | 0 | 0 | 5
  Scattered Areas of Fibroglandular Density | 196 | 20 | 4 | 220
  Heterogeneously Dense | 140 | 13 | 10 | 163
  Extremely Dense | 11 | 2 | 0 | 13
  Unknown | 5 | 0 | 0 | 5
Palpability [Count of Participants; unit: Participants]
  Palpable Mass | 85 | 11 | 4 | 100
  Not palpable Mass | 272 | 24 | 10 | 306
Tumor Histology From Biopsy [Count of Participants; unit: Participants]
  DCIS only | 70 | 6 | 2 | 78
  IDC +/- DCIS | 249 | 25 | 10 | 284
  ILC +/- DCIS | 35 | 4 | 2 | 41
  IDC + ILC | 3 | 0 | 0 | 3
Estrogen Receptor (ER) (+) Genetic Marker from Biopsy [Count of Participants; unit: Participants]
  ER (+) | 335 | 30 | 13 | 378
  ER (-) | 19 | 5 | 1 | 25
  Not available | 3 | 0 | 0 | 3
Progesterone Receptor (PR) (+) Genetic Marker from Biopsy [Count of Participants; unit: Participants]
  PR (+) | 272 | 28 | 11 | 311
  PR (-) | 48 | 5 | 1 | 54
  Unknown | 37 | 2 | 2 | 41
Human Epidermal growth factor Receptor 2 (HER2) (+) Genetic Marker from Biopsy [Count of Participants; unit: Participants]
  HER2 (+) | 20 | 3 | 0 | 23
  HER2 (-) | 280 | 26 | 13 | 319
  Unknown | 57 | 6 | 1 | 64
Triple Negatives Genetic Marker from Biopsy [Count of Participants; unit: Participants]
  Triple Negatives - Yes | 11 | 3 | 1 | 15
  Triple Negatives - No | 346 | 32 | 13 | 391
Lymph Nodes Biopsy [Count of Participants; unit: Participants]
  Lymph Node (+) | 9 | 1 | 0 | 10
  Lymph Node (-) | 51 | 7 | 2 | 60
  No Lymph Node Biopsy | 297 | 27 | 12 | 336

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Had Residual Cancer Found in at Least One LUM Imaging System Guided Shave Among All Patients.
Description: Residual cancer was defined as tumor found by pathology in a therapeutic shave after the SOC surgical procedure was completed; that is, tumor that current Standard of Care (SOC) surgery failed to remove. LUM Imaging System was used during the surgery, but the assessment of the outcomes was unknown until the pathology report was available.
Time Frame: Day 1, during surgery
Population: modified intent to treat population (mITT) includes subjects injected with LUM015 and LUM Imaging was performed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Device Intervention: LUM Imaging System Used: The LUM Imaging Device was used to examine inside the lumpectomy cavity to determine if the dye indicated any areas that might contain residual tumor. If the imaging tested positive for the cancer cells remaining in the lumpectomy cavity, the surgeon would remove an additional piece of tissue. This process was continued until a negative reading from the device was obtained or a maximum of 2 shaves of additional tissue had been removed. Patients in this arm received the study drug, LUM015.
  Study Device Arm: LUM015 was administered 2 to 6 hours prior to surgery. The LUM Imaging device was used to assist in the removal of additional tumor tissue.
Arm/Group | Device Intervention: LUM Imaging System Used
Number analyzed (Participants) | 357
percentage of participants | 7.6 [5.0 to 10.8]

2. Primary Outcome: Sensitivity of LUM Imaging System on Cancer in the Lumpectomy Cavity
Description: Sensitivity of LUM Imaging System on cancer was calculated as percentage of tissues with cancer that was removed from lumpectomy cavity due to positive detection by LUM Imaging System. The estimates of the instrument diagnostic sensitivity used Generalized Estimating Equations (GEE) approach. This method was used to analyze correlated data which was modeled with generalized linear model having binomial link function and including correlation cluster and matrix information (here within each subject). LUM Imaging System was used during the surgery, but the assessment of the outcomes was unknown until the pathology report was available.
Time Frame: Day 1, during surgery
Population: modified intent to treat population (mITT) includes subjects injected with LUM015 and LUM Imaging was performed
Measure: Number (95% Confidence Interval); unit: percentage of tissues with cancer
Units Other Than Participants: Tissue with cancer
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery
Number analyzed (Participants) | 357
Number analyzed (Tissue with cancer) | 69
percentage of tissues with cancer | 49.1 [36.4 to 61.9]

3. Secondary Outcome: Detection and Conversion of Positive Margins.
Description: Detection of positive margins: Percentage of patients with positive margins after standard of care breast-conserving surgery, all had LUM Imaging System signals above the threshold in the cavity as defined by the tumor detection algorithm.
  Conversion of positive margins: Percentage of patients with positive margins after standard of care breast-conserving surgery resulted in the negative margin after LUM Imaging System was used.
  The system was used during the surgery, but the assessment of the outcomes was unknown until the pathology report was available.
Time Frame: Day 1, during surgery
Population: modified intent to treat population (mITT) includes subjects injected with LUM015 and LUM Imaging was performed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery
Number analyzed (Participants) | 357
percentage of participants
  Percentage among participants having positive margins after SoC all detected by LUM Imaging System: number analyzed (Participants) | 62
  Percentage among participants having positive margins after SoC all detected by LUM Imaging System | 16.1 [8.0 to 27.7]
  Percentage of participants with positive SOC margins converted to negative with LUM Imaging System: number analyzed (Participants) | 62
  Percentage of participants with positive SOC margins converted to negative with LUM Imaging System | 14.5 [6.9 to 25.8]

4. Secondary Outcome: Removal of Residual Cancer Guided by the LUM Imaging System in Participants With Negative Margins After Standard-of-Care Surgery
Description: Percentage of participants having residual tumor removed within subpopulation of having negative margins after Standard of Care surgery. The system was used during the surgery, but the assessment of the outcomes was unknown until the pathology report was available.
Time Frame: Day 1, during surgery
Population: Participants having negative margin after standard of care procedure of lumpectomy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery
Number analyzed (Participants) | 295
percentage of participants | 6.4 [3.9 to 9.9]

5. Secondary Outcome: Removal of Residual Cancer Guided by the LUM Imaging System in Subjects With Positive Margins After Standard-of-Care Surgery
Description: Percentage of participants having residual tumor removed within subpopulation of having positive margins after Standard of Care surgery. The system was used during the surgery, but the assessment of the outcomes was unknown until the pathology report was available.
Time Frame: Day 1, during surgery
Population: Participants with positive margins after standard of care procedure of lumpectomy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery
Number analyzed (Participants) | 62
percentage of participants | 12.9 [5.7 to 23.9]

6. Secondary Outcome: Volume of Therapeutic Shaves Removed During Lumpectomy.
Description: The median volumes of Lumicell Imaging System - guided shaves (therapeutic shaves) were measured and the median total volume removed during lumpectomy was presented as well. The system was used during the surgery, but the assessment of the outcomes was unknown until the pathology report was available.
Time Frame: Day 1, during surgery
Population: mITT and control populations
Measure: Median (95% Confidence Interval); unit: cm^3
Groups:
- Standard of Care Arm: The LUM Imaging Device was not used to guide additional tissue removal. Patients in this arm will receive the study drug, LUM015.
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery | Standard of Care Arm
Number analyzed (Participants) | 357 | 35
cm^3
  Lumpectomy volume | 54 [9.7 to 267.2] | 66.8 [10.5 to 308.0]
  SOC shave volume | 7.5 [0 to 71.2] | 7.7 [0 to 71.9]
  SOC total volume | 66.4 [15.1 to 308.7] | 76.7 [21.9 to 308]
  Therapeutic shave volume | 0 [0 to 61.1] | 0 [0 to 0]
  Total volume | 77.5 [15.2 to 348.1] | 76.7 [21.9 to 308.0]

7. Secondary Outcome: Contribution of Therapeutic Shaves to Total Volume Removed During Lumpectomy.
Description: Median of the percentages of the volumes of Lumicell Imaging System - guided shaves (therapeutic shaves) out of total volume removed during lumpectomy for each participant were measured. The system was used during the surgery, but the assessment of the outcomes was unknown until the pathology report was available.
Time Frame: Day 1, during surgery
Population: mITT and Control arm populations
Measure: Median (95% Confidence Interval); unit: Percent
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery | Standard of Care Arm
Number analyzed (Participants) | 357 | 35
Percent | 0 [0 to 44.7] | 0 [0 to 0]

8. Primary Outcome: Specificity of LUM Imaging System Detection on Cancer in the Lumpectomy Cavity
Description: Specificity of LUM Imaging System Detection on Cancer in the Lumpectomy Cavity was measured as percentage of the negative margins without cancer, that were tested negative by LUM Imaging System. The estimate of the instrument diagnostic specificity used Generalized Estimating Equations (GEE) approach with random effects from intraclass correlation within subjects.
Time Frame: Day 1, during surgery
Population: modified intent to treat population (mITT) includes subjects injected with LUM015 and LUM Imaging was performed
Measure: Number (95% Confidence Interval); unit: percentage of negative margins w/o ca
Units Other Than Participants: Negative margins without cancer
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery
Number analyzed (Participants) | 357
Number analyzed (Negative margins without cancer) | 2277
percentage of negative margins w/o ca | 86.5 [84.5 to 88.3]

ADVERSE EVENTS:
Time Frame: All adverse events and adverse device effects, both serious and non-serious, and deaths that are encountered from initiation of study intervention, throughout the study, and within the first post-operative follow-up visit should be followed to their resolution, or until the principal investigator assesses them as stable, or the principal investigator determines the event to be irreversible, or the subject is lost to follow-up. Adverse events were assessed up to 30 days after enrollment.
Description: Serious adverse events should be reported within 24 hours of learning of the occurrence. Non-serious adverse events and non-serious adverse device effects will be reported to Lumicell on the adverse events Case Report Forms during the study.
Arm/Group | Device Intervention: LUM Imaging System Used During Surgery | Standard of Care Arm | Withdrawn Before Randomization
All-Cause Mortality (participants affected / at risk) | 0/357 | 0/35 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/357 | 0/35 | 2/14
Other Adverse Events (participants affected / at risk) | 334/357 | 32/35 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Intervention: LUM Imaging System Used During Surgery (N=357) | Standard of Care Arm (N=35) | Withdrawn Before Randomization (N=14)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Intervention: LUM Imaging System Used During Surgery (N=357) | Standard of Care Arm (N=35) | Withdrawn Before Randomization (N=14)
Chromaturia (Renal and urinary disorders) | 325 (325) | 30 (30) | 13 (13)
Breast pain (Reproductive system and breast disorders) | 20 (22) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 11 (11) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 10 (10) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Extravasation (General disorders) | 1 (2) | 0 (0) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 22 (22) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Our trial did not take additional margin specimens from cavity orientations with negative Pegulicianine fluorescence-guided (pFGS) readings but scored the pFGS cavity reading as falsely negative if the corresponding lumpectomy margin was positive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT03686215/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03686215/SAP_001.pdf